CLINICAL TRIAL: NCT00684606
Title: Transcervical Foley Catheter With or Without IV Oxytocin Infusion for Induction of Labor: a Randomized Controlled Trial
Brief Title: Transcervical Foley Catheter With or Without Oxytocin for Induction of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Orit Moran, Sheba Medical Cener
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-08-5164-OM-CTIL
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Pregnancy; Induction of Labor
Keywords: Induction of Labor; Low Bishop Score; Transcervical Foley Catheter.; IV Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Transcervical Foley catheter with IV Oxytocin
  Interventions: Drug: Oxytocin IV
- 2 (No Intervention): Transcervical Foley catheter only

INTERVENTIONS:
Drug: Oxytocin IV — 5 miu/1000ml Glu/Saline
  Other Names: Pitocin
  Arms: 1

SUMMARY:
The purpose of the present study is to evaluate the possible benefit of concurrent IV Oxytocin infusion with trans cervical Foley catheter for pre-induction cervical ripening.

DETAILED DESCRIPTION:
Induction of labor in term pregnancy may be challenging, especially in patients with unfavorable cervical conditions. Numerous trails have presented evidence of the efficacy of the trans cervical Foley catheter for pre-induction cervical ripening.The purpose of the present study is to evaluate the possible benefit of concurrent IV Oxytocin infusion with trans cervical Foley catheter for pre-induction cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Medical indication for labor induction by transcervical Foley catheter

Exclusion Criteria:

* Preterm pregnancy
* Contraindication for induction of labor by transcervical Foley catheter or by IV Oxytocin:

  * Uterine scar
  * Multiple pregnancy
  * PROM
  * Grand-multiparity
  * Placenta previa or marginal placenta
  * Spontaneous uterine contractions (more than 3 in 10 minutes)
  * Vaginal bleeding
  * Nonreassuring fetal heart rate

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The period of time needed for ripening the uterine cervix by Transcervical Foley catheter with or without IV Oxytocin infusion. | year

CONTACTS AND LOCATIONS:
Overall Officials: Orit Moran, M.D., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel